CLINICAL TRIAL: NCT00278018
Title: Peritumoral Injection of Immature Dendritic Cels to Irradiated Metastases of Solid Tumors
Brief Title: Peritumoral Injection of Immature Dendritic Cells to Irradiated Skin Metastases of Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Because there were no responses
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: immatureDC- HMO-CTIL
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2007-04

CONDITIONS: Cancer of Skin; Solid Tumors
MeSH Terms: conditions — Skin Neoplasms

INTERVENTIONS:
Procedure: Immunotherapy treatment for solid tumors

SUMMARY:
Melanoma is the main cause of death in patients with skin cancer. Once it has metastasized, this cancer has been shown to respond to chemotherapy only in rare cases. Immunotherapy represents an approach to treatment based on the immune response to cancer antigens.

The long-term objective of this study is to develop a therapeutic approach for the treatment of cancer in general, and melanoma in particular, based on immunotherapy, using a combination of local tumor irradiation followed by injection of immature dendritic cells (iDC).The treatment will be followed by the injection of interferon alpha, which we expect will induce activation of the iDC.

This trial is based on the hypothesis that local radiation, which causes destruction of the tumor, in combination with injection of the patient's own iDC and the activation of these cells with interferon alpha, will induce an effective immune response against the tumor. In order to test the suggested approach, we propose a 20-patients clinical trial that will evaluate the objective clinical and immunological response to the proposed treatment in patients with malignant melanoma and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient above age 18, with measurable metastatic melanoma or other solid tumor, with at least one tumor deposit that is easily accessible to peri-tumoral DC injection. The preferred location is subcutaneous or intradermal. Patients with additional metastatic sites will not be excluded. Patients should have an expected survival of greater than three months.

   Patient must have received accepted standard treatment of his or her cancer:
   * for melanoma - DTIC -containing protocol ,unless unwilling. Previous treatment with IL-2 is not an excluding factor.
   * for breast cancer - adriamycin and cyclophosphamide, taxanes, and vinorelbine-containing protocols
   * for lung, renal and GIT cancers- one previous chemotherapy line
2. Serum creatinine of 2.0 mg/dl or less.
3. Total bilirubin 1.6 mg/dl or less, except for patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
4. WBC 3000/mm3 or greater.
5. Platelet count 90,000 mm3 or greater.
6. Serum AST/ALT less then two times normal.
7. ECOG performance status of 0, 1 or 2.
8. Patients of both genders must be willing to practice effective birth control during this trial.
9. Patient agreed to participate in the study and has signed a written informed consent.

Exclusion Criteria:

Patients will be excluded:

1. who are undergoing or have undergone in the past 3 weeks any other form of therapy except from surgery for their cancer.
2. have active systemic infections, coagulation disorders, autoimmune disease or other major medical illnesses of the cardiovascular or respiratory systems or any known immunodeficiency disease.
3. who require steroid therapy.
4. who are pregnant (because of possible side effects on the fetus).
5. who are known to be positive for hepatitis B and C or HIV antibody (because of possible immune effects of these conditions).
6. who have any form of primary or secondary immunodeficiency. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
7. who are allergic to eggs.

i. who have an active major medical illnesses such as cardiac ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Complete evaluation of untreated lesions with physical examination and appropriate X-rays and/or scans will be performed four to six weeks after the last DC injection.
Immunological evaluation will be performed two weeks after the last DC injection.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Lotem, MD, Principal Investigator — Hadassah Medical Organization, pob 12000, Jerusalem, Israel
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel